CLINICAL TRIAL: NCT05056831
Title: Efficacy of an Adapted Multicomponent Physical Activity Intervention to Reduce Psychosocial Distress in Rural Adults Following Cancer Diagnosis
Brief Title: Multicomponent Physical Activity Intervention for the Reduction of Psychosocial Distress in Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Kawut, Steven, MD (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1278; NCI-2021-09572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1278 (Other: M D Anderson Cancer Center); K07CA222335 (NIH); R01HL142732 (NIH)
Record Dates: First submitted 2021-08-25; First posted 2021-09-27 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Anxiety Disorder; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Anxiety Disorders; Hematologic Neoplasms | interventions — Behavior Therapy; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (physical activity intervention) (Experimental): Patients attend face-to-face mind-body sessions focused on stretching, breathing, and relaxation twice a week and receive targeted text messages daily on their smartphone for 8 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (usual care) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Attend face-to-face mind-body sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Group I (physical activity intervention)
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group II (usual care)
Other: Informational Intervention — Receive targeted text messages
  Arms: Group I (physical activity intervention)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study adapts and assesses the effect of a multicomponent physical activity intervention in reducing psychosocial distress in cancer patients. This study aims to develop a program to help increase physical activity and reduce stress in cancer survivors who live in rural areas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To adapt a multicomponent intervention (HH+AIM) that assesses the perspective of health care provider and cancer survivors about:

Ia. Needs related to psychosocial distress and health behaviors in rural patients with cancer.

Ib. Needs related to implementing interventions within the treatment setting. Ic. Barriers to intervention delivery/participate. Id. Preferred means/methods for referring participants and receiving information related to the intervention.

SECONDARY OBJECTIVES:

I. To assess time spent sitting in prolonged bouts of 20 consecutive minutes or more (minutes/day).

II. To assess daily number of steps (collected using the activPAL over 7 days at week 8, data will be averaging over 7 days to get minutes per day).

III. To assess psychosocial distress measured using the National Comprehensive Cancer Network (NCCN) Distress Thermometer scores.

IV. To assess health-related quality of life measured using the SF-36 short form.

OUTLINE:

PART I: Patients and providers complete a questionnaire and attend an interview over 1 hour.

PART II: Patients are randomized to 1 of 2 groups.

GROUP I: Patients attend face-to-face mind-body sessions focused on stretching, breathing, and relaxation twice a week and receive targeted text messages daily on their smartphone for 8 weeks.

GROUP II: Patients receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* PROVIDERS: Work with cancer survivors (e.g., radiation and medical oncologists, oncology nurses, oncology patient navigators, and clinical research coordinators)
* PROVIDERS: Place of engagement falls within a rural county in Texas
* PROVIDERS: Able to read, speak, and write in English
* PROVIDERS: At least 18 years old
* PROVIDERS: Have access to a smartphone, tablet, or computer with internet access and willing to attend virtual sessions
* INTERVIEW SURVIVORS: Men and women >= 18 years of age
* INTERVIEW SURVIVORS: History of cancer
* INTERVIEW SURVIVORS: Currently receiving treatment or have recently completed treatment but are still attending appointments at UTHealth North Campus Tyler (=< 1 year)
* INTERVIEW SURVIVORS: Able to read, speak, and write in English
* INTERVIEW SURVIVORS: Have access to a smartphone, tablet, or computer with internet access and willing to attend virtual sessions
* INTERVENTION SURVIVORS: Men and women >= 18 years of age
* INTERVENTION SURVIVORS: Received a solid tumor cancer diagnosis stage I-III
* INTERVENTION SURVIVORS: Receiving radiation therapy or planning to receive radiation therapy for a solid tumor diagnosis for at least 4 weeks
* INTERVENTION SURVIVORS: Able to engage in moderate intensity physical activity as determined by the Physical Activity Readiness Questionnaire (PAR-Q) or by physicians clearance (letter from physician or nurse practitioner)
* INTERVENTION SURVIVORS: Physician clearance to participate in the study
* INTERVENTION SURVIVORS: Physically inactive (=< 60 minutes of moderate or greater physical activity [PA] per week during the past 6 months)
* INTERVENTION SURVIVORS: Live within MD Anderson's rural catchment area
* INTERVENTION SURVIVORS: Have a home address where information can be mailed and a working telephone
* INTERVENTION SURVIVORS: Have access to a smartphone, tablet, or computer with internet access and willing to attend virtual sessions
* INTERVENTION SURVIVORS: Able to read, speak, and write in English
* INTERVENTION SURVIVORS: Able to receive text messages on their smartphone (via cellular data or wireless internet)

Exclusion Criteria:

* PROVIDERS: Does not work with cancer survivors
* PROVIDERS: Place of work or engagement falls within an urban/metropolitan county in Texas
* PROVIDERS: Does not read, speak, or write in English
* PROVIDERS: Below the age of 18 years
* INTERVIEW SURVIVORS: No history of cancer
* INTERVIEW SURVIVORS: Does not read, speak, or write in English
* INTERVIEW SURVIVORS: Below the age of 18
* INTERVENTION SURVIVORS: No history of cancer
* INTERVENTION SURVIVORS: Have absolute contraindications to unassisted physical activity (e.g., acute myocardial infarction, severe orthopedic or musculoskeletal limitations)
* INTERVENTION SURVIVORS: Currently participating in another intervention to increase physical activity or reduce sedentary behavior
* INTERVENTION SURVIVORS: Self-report meeting physical activity recommendations (>= 60 minutes of moderate or greater PA per week during the past 6 months)
* INTERVENTION SURVIVORS: Physical limitations that might be aggravated by participation in moderate-intensity physical activity as measured using the Physical Activity Readiness Questionnaire (PAR-Q), and any physical limitation that prevents engaging in moderate intensity exercise
* INTERVENTION SURVIVORS: Primary address falls within an urban/metropolitan county in Texas
* INTERVENTION SURVIVORS: Plan to move from the area or discontinue their treatment at UTHealth North Campus Tyler during the 14-week study period
* INTERVETION SURVIVORS: Does not read, speak, or write in English
* INTERVENTION SURVIVORS: Below the age of 18
* INTERVENTION SURVIVORS: Pregnant or planning to become pregnant during the 14 week study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
To establish a multicomponent intervention that assesses the perspective of health care provider | Through study completion, an average of 1 year
To establish a multicomponent intervention that assesses the perspective of cancer survivors | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Scherezade Mama, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT05056831/ICF_000.pdf